CLINICAL TRIAL: NCT03578952
Title: Evaluation of Effectiveness and Safety of Evolut R Valve In Patients With Pure Aortic Regurgitation Transcatheter Aortic Valve Replacement for Pure Severe Aortic Regurgitation Pilot Study
Brief Title: Evaluation of Effectiveness and Safety of Evolut R Valve In Patients With Pure Aortic Regurgitation
Acronym: Pure AR TAVR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of support
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Department of Medicine, Heart Institute, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2018-06
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve; Aortic Valve Insufficiency; Aortic Regurgitation; Regurgitation, Aortic Valve; Aortic Incompetence
Keywords: TAVR; TAVI; Pure AR
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pure AR (Experimental): Patients with symptomatic severe aortic valve regurgitation without severe aortic stenosis requiring aortic valve replacement.
  Interventions: Device: TAVR with Evolut R valve

INTERVENTIONS:
Device: TAVR with Evolut R valve — TAVR with Evolut R valve

SUMMARY:
This study is to evaluate the efficacy and safety of transcatheter aortic valve replacement (TAVR) in severe 'pure Aortic regurgitation (AR)' using Evolut R valve (Medtronic, Minneapolis, MN).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have co-morbidities such that the principal investigator and co-investigator concur that the predicted risk of operative mortality is ≥15% (STS score ≥10 OR Logistic EuroSCORE ≥20%).

   A candidate who does not meet [the STS score criteria ≥ 10 OR Logistic EuroSCORE ≥20%] can be included in the study if a peer review by at least two investigators concluded and documented that the patient's predicted risk of operative mortality is ≥15% from old age, severe frailty or STS score ≥8. In this case, all evidence must be documented in the study case report form as well as in the patient medical record.
2. There is a formal agreement by a cardiac surgeon, echo part cardiologist and interventional cardiologist according to the relevant guideline.
3. The subject does not have severe degenerative aortic stenosis and do have severe aortic regurgitation.
4. The subject or the subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
5. The subject agrees that the subject will keep in touch with study team for all required post-procedures like angiography or transesophageal echography.
6. The subject agrees that the subject will cooperate with study team for all required post-procedure visits.
7. The subject's age is 20 or more.

Exclusion Criteria:

1. Evidence of an acute myocardial infarction ≤ 1 month before the intended treatment(defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition).
2. Any therapeutic invasive cardiac procedure performed within 30 days of the index procedure, (or 6 months if the procedure was a drug-eluting coronary stent implantation).
3. Blood dyscrasias as defined: leukopenia (WBC<3000 mm3), acute anemia (Hb<9 mg%), thrombocytopenia (platelet count <50,000 cells/mm³), history of bleeding diathesis or coagulopathy.
4. Untreated clinically significant coronary artery disease requiring revascularization.
5. Need for emergency surgery for any reason.
6. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
7. Active bacterial endocarditis or other active infections.
8. Active peptic ulcer or upper GI bleeding within the prior 3 months.
9. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine (Ticlid), or clopidogrel (Plavix), or sensitivity to contrast media, which cannot be adequately pre-medicated.
10. Recent (within 6 months) cerebrovascular accident (CVA) or a transient ischemic attack (TIA).
11. Life expectancy < 12 months due to non-cardiac comorbid conditions.
12. Significant aortic disease, including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5cm or greater; marked tortuosity (hyperacute bend or angle of aortic arch ≥200 degree),aortic arch atheroma (especially if thick [> 5mm], protruding or ulcerated) or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta (applicable for transfemoral patients only).
13. Root disease including annuloaortic ectasia or aneurysm of root or sinus.
14. Iliofemoral vessel characteristics that would preclude safe placement of introducer sheath such as severe obstructive calcification, severe tortuosity(with moderate or severe calcification and two or more severe curve (angle ≥90°) (applicable for transfemoral patients only).
15. Pregnant(positive result from pregnancy test conducted during screening visit and within prior 2 weeks of valve replacement) or lactating women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Aortic regurgitation | 1 month

SECONDARY OUTCOMES:
All cause death | 1 month, 6 months, 1,2,3 and 5 years
Cardiovascular mortality | 1 month, 6 months, 1,2,3 and 5 years
Stroke | 1 month, 6 months, 1,2,3 and 5 years
  Valve Academic Research Consortium (VARC)
Myocardial Infarction | 1 month, 6 months, 1,2,3 and 5 years
  Valve Academic Research Consortium (VARC)
Re-hospitalization | 1 month, 6 months, 1,2,3 and 5 years
Acute kidney injury | 7 days
  Valve Academic Research Consortium (VARC)
Vascular access site and access-related complication | 7 days
  Valve Academic Research Consortium (VARC)
Bleeding | 7 days
  Valve Academic Research Consortium (VARC)
Acute kidney injury | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided